CLINICAL TRIAL: NCT02904590
Title: A Prospective Study on the Incidence and Risk Factors Related to Infection in Patients With Inflammatory Bowel Disease
Acronym: INFEII
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Other Study IDs: INFEII
Record Dates: First submitted 2016-08-26; First posted 2016-09-19 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; Infection
MeSH Terms: conditions — Inflammatory Bowel Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood sample of 10 cc
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IBD patients: Incidental patients with IBD controlled (including Crohn's disease, Ulcerative colitis and unclassified colitis)

SUMMARY:
The purpose of this study is to determine the incidence and risk factors related to Infection in patients with Inflammatory Bowel Disease (IBD)

DETAILED DESCRIPTION:
IBD could lead to an increased risk of infections, particularly related to immunosuppressive therapy. The true effect of having IBD in the development of infections has not been studied in depth since the cohort studies are scarce and the results of studies with different approaches are contradictory.

The limited time period of former studies may not be enough to assess infectious complications that may occur in a long term period.

Moreover, certain polymorphisms demonstrated to confer a higher risk of opportunistic infections under immunosuppressive conditions, for instance HIV, patients with cystic fibrosis and Candida' infections. For this reason, it seems reasonable to think that genetic factors might play a role in the risk of opportunistic infections in IBD.

The hypothesis of this study is that patients with IBD have an increased risk of infection by immunosuppressive treatment.

TYPE OF STUDY Prospective cohort study that evaluates the effect of immunosuppression and other clinical factors in the onset of infection in IBD

STUDY DESIGN PATIENTS & METHODS This study is aimed to all incidental patients diagnosed with Crohn's disease and ulcerative colitis included in the ENEIDA database.

METHODS An infection would be considered as relevant when: 1) requires hospital admission, 2) leads to death or endangers the patient's life (ICU admission, presence of hemodynamic instability, sepsis, tracheal intubation, vasoactive drug requirement), 3) must be treated with specific antibiotics (antibacterials, antivirals, antifungals) 4) affects recurrently (herpes virus, papilloma virus, etc). 5) requires change/withdrawal of immunosuppressive or biological treatment.

The appearance of relevant infection will be prospectively evaluated, performing a subanalysis at 3 and 5 years using ENEIDA platform. ENEIDA is a database from a Spanish national study in IBD on genetic and environmental determinants run under GETECCU (Grupo Español de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa) supervision. This database basically comprises: demographic characteristics, type of IBD, immunosuppressant treatment, biological treatment or surgery)

At the time of inclusion the following variables should be available (and are mandatory): demographic characteristics, type of IBD, date of diagnosis, phenotypic characteristics of the disease, history of serious infections, information on received treatments particularly the exposure to immunosuppressants, biological treatment or surgery and whether an infection has occurred as a complication of the three treatment groups. It should also be collected the following serologic details: hepatitis type B virus C, HIV, tuberculosis (TB), varicella zoster status.

At the time of registration a blood sample (10cc) will be drawn and sent to a biobank to analyze the DNA for genetic research.

STUDY ANALYSIS Sample calculation

The main objective of this study is to determine the percentage of infections in IBD and the related risk factors for the development of infections in patients with IBD. Given that the reported prevalence of infection varies between 6 and 10%the formula for estimating endless samples, establishing:

* Security level of the confidence interval at 95%
* Expected value for the worst case scenario of 6% (prevalence of infection)
* Precision of 1.5%
* The minimum sample number is set to 963, and assuming a loss rate of 20%

With these assumptions, the total number of patients to be included is 1204 patients.

The statistical analysis will be in three steps: (1) independent clinical factors analysis, (2) genetic factors infection-related analysis and (3) clinical and genetic factors infection- related analysis.

Baseline and follow up data will be compared among patients who develop infection and those who do not. Quantitative variables will be contrast by T-student and Mann-Whitney test. Qualitative variable will be contrast by X2 or Fisher test. Logistic regression will be conducted to analyze independent associations between variables and Kaplan-Meier test to calculate survival curves.

An analysis of Cox proportional hazards will be conducted to assess the effect of exposure to independent predictors of the risk of significant infection or mortality.

Finally the intensity of the significant associations will be measured by calculating the OR, HR and confidence interval of 95%.

ELIGIBILITY:
Inclusion criteria:

* All incidental patients with IBD controlled at each participating center, registered in the ENEIDA database could be included, until the expected study sample is reached (n=1204 patients).
* An incidental IBD case is any patient with a diagnosis of Crohn's disease, ulcerative colitis and unclassified colitis after 3-6 month of the conclusive diagnosis of IBD.

Exclusion Criteria:

* HIV infection or any congenital immunodeficiency at the time of inclusion.
* To be under any immunosuppressant therapy for another reason other than IBD at IBD diagnosis.
* No consent to participate.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Incident cases of IBD registered on ENEIDA data base
Sampling Method: Probability Sample
Enrollment: 1204 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
The incidence of infection and type of infection in patients with ulcerative colitis and Crohn's disease, regardless of treatment received. ulcerative colitis and Crohn's disease, regardless of treatment received. | Change from baseline incidence and type of infection at 3 and 5 years
  Serious infection means any untoward medical occurrence that at any dose:
  * Results in death or life-threatening
  * Requires in patient hospitalization or prolongation of an existing hospitalization
  * Is a medically important event.
  * Requires specific chemotherapy treatment
  * Emerges repeatedly.
  * Induces a switch or a withdrawal of the immunosuppressive or biological treatment
Clinical, demographic, epidemiologic and genetic factors associated with the risk of infection in patients with IBDassociated with the risk of infection in patients with IBD. | Change from baseline and at 3 and 5 years

SECONDARY OUTCOMES:
The effect of duration and immunosuppressive potency in the development of infections | at baseline and at 3 and 5 years
The impact of infection on morbidity and mortality in patients with IBD. | at baseline and at 3 and 5 years
The type of infections in IBD patients grouped by systems and whether they are opportunistic or not. | at baseline and at 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yamile Zabana, Principal Investigator — Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa
Locations (24):
- Spain (24):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Althaia, xarxa assistencial universitaria de Manresa, Manresa, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de Galdakao, Galdakao, Bilbao
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital General de Tomelloso, Tomelloso, Ciudad REAL
  - Hospital Universitario Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Complexo Hospital Universitario de Vigo, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital De La Princesa, Madrid
  - Consorci hospitalari de Terrassa, Terrassa
  - Hospital Clínic de València, Valencia
  - Hospital Universitari La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford AC, Peyrin-Biroulet L. Opportunistic infections with anti-tumor necrosis factor-alpha therapy in inflammatory bowel disease: meta-analysis of randomized controlled trials. Am J Gastroenterol. 2013 Aug;108(8):1268-76. doi: 10.1038/ajg.2013.138. Epub 2013 May 7. PMID 23649185
- [Background] Toruner M, Loftus EV Jr, Harmsen WS, Zinsmeister AR, Orenstein R, Sandborn WJ, Colombel JF, Egan LJ. Risk factors for opportunistic infections in patients with inflammatory bowel disease. Gastroenterology. 2008 Apr;134(4):929-36. doi: 10.1053/j.gastro.2008.01.012. Epub 2008 Jan 11. PMID 18294633
- [Background] Lichtenstein GR, Feagan BG, Cohen RD, Salzberg BA, Diamond RH, Chen DM, Pritchard ML, Sandborn WJ. Serious infections and mortality in association with therapies for Crohn's disease: TREAT registry. Clin Gastroenterol Hepatol. 2006 May;4(5):621-30. doi: 10.1016/j.cgh.2006.03.002. PMID 16678077
- [Background] Lichtenstein GR, Feagan BG, Cohen RD, Salzberg BA, Diamond RH, Price S, Langholff W, Londhe A, Sandborn WJ. Serious infection and mortality in patients with Crohn's disease: more than 5 years of follow-up in the TREAT registry. Am J Gastroenterol. 2012 Sep;107(9):1409-22. doi: 10.1038/ajg.2012.218. Epub 2012 Aug 14. PMID 22890223
- [Background] Beaugerie L, Gerbes AL. Liver dysfunction in patients with IBD under immunosuppressive treatment: do we need to fear? Gut. 2010 Oct;59(10):1310-1. doi: 10.1136/gut.2010.217331. No abstract available. PMID 20833661
- [Background] Papadopoulos AI, Ferwerda B, Antoniadou A, Sakka V, Galani L, Kavatha D, Panagopoulos P, Poulakou G, Protopapas K, van der Meer JW, Netea MG, Giamarellos-Bourboulis EJ. Association of Mal/TIRAP S180L variant polymorphism with decreased infection risk in patients with advanced HIV-1 infection. Cytokine. 2012 Oct;60(1):104-7. doi: 10.1016/j.cyto.2012.05.008. Epub 2012 Jun 8. PMID 22683004
- [Background] Radovanovic I, Mullick A, Gros P. Genetic control of susceptibility to infection with Candida albicans in mice. PLoS One. 2011 Apr 20;6(4):e18957. doi: 10.1371/journal.pone.0018957. PMID 21533108
- [Background] Papadopoulos AI, Ferwerda B, Antoniadou A, Sakka V, Galani L, Kavatha D, Panagopoulos P, Poulakou G, Kanellakopoulou K, van der Meer JW, Giamarellos-Bourboulis EJ, Netea MG. Association of toll-like receptor 4 Asp299Gly and Thr399Ile polymorphisms with increased infection risk in patients with advanced HIV-1 infection. Clin Infect Dis. 2010 Jul 15;51(2):242-7. doi: 10.1086/653607. PMID 20521908
- [Background] Pine SO, McElrath MJ, Bochud PY. Polymorphisms in toll-like receptor 4 and toll-like receptor 9 influence viral load in a seroincident cohort of HIV-1-infected individuals. AIDS. 2009 Nov 27;23(18):2387-95. doi: 10.1097/QAD.0b013e328330b489. PMID 19855253
- [Background] Jurevic RJ, Bai M, Chadwick RB, White TC, Dale BA. Single-nucleotide polymorphisms (SNPs) in human beta-defensin 1: high-throughput SNP assays and association with Candida carriage in type I diabetics and nondiabetic controls. J Clin Microbiol. 2003 Jan;41(1):90-6. doi: 10.1128/JCM.41.1.90-96.2003. PMID 12517831
- [Background] Connelly TM, Sehgal R, Berg AS, Hegarty JP, Deiling S, Stewart DB, Poritz LS, Koltun WA. Mutation in TAGAP is protective of anal sepsis in ileocolic Crohn's disease. Dis Colon Rectum. 2012 Nov;55(11):1145-52. doi: 10.1097/DCR.0b013e3182676931. PMID 23044675
- [Background] Obrador A, Lopez San Roman A, Munoz P, Fortun J, Gassull MA; Grupo Espanol de Trabajo de Enfermedad de Crohn y Colitis Ulcerosa (GETECCU). [Consensus guideline on tuberculosis and treatment of inflammatory bowel disease with infliximab. Spanish Working Group on Crohn Disease and Ulcerative Colitis]. Gastroenterol Hepatol. 2003 Jan;26(1):29-33. doi: 10.1016/s0210-5705(03)70338-0. No abstract available. Spanish. PMID 12525326
- [Background] Arts J, D'Haens G, Zeegers M, Van Assche G, Hiele M, D'Hoore A, Penninckx F, Vermeire S, Rutgeerts P. Long-term outcome of treatment with intravenous cyclosporin in patients with severe ulcerative colitis. Inflamm Bowel Dis. 2004 Mar;10(2):73-8. doi: 10.1097/00054725-200403000-00002. PMID 15168804
- [Background] Fidder H, Schnitzler F, Ferrante M, Noman M, Katsanos K, Segaert S, Henckaerts L, Van Assche G, Vermeire S, Rutgeerts P. Long-term safety of infliximab for the treatment of inflammatory bowel disease: a single-centre cohort study. Gut. 2009 Apr;58(4):501-8. doi: 10.1136/gut.2008.163642. Epub 2008 Oct 2. PMID 18832524
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Jostins L, Ripke S, Weersma RK, Duerr RH, McGovern DP, Hui KY, Lee JC, Schumm LP, Sharma Y, Anderson CA, Essers J, Mitrovic M, Ning K, Cleynen I, Theatre E, Spain SL, Raychaudhuri S, Goyette P, Wei Z, Abraham C, Achkar JP, Ahmad T, Amininejad L, Ananthakrishnan AN, Andersen V, Andrews JM, Baidoo L, Balschun T, Bampton PA, Bitton A, Boucher G, Brand S, Buning C, Cohain A, Cichon S, D'Amato M, De Jong D, Devaney KL, Dubinsky M, Edwards C, Ellinghaus D, Ferguson LR, Franchimont D, Fransen K, Gearry R, Georges M, Gieger C, Glas J, Haritunians T, Hart A, Hawkey C, Hedl M, Hu X, Karlsen TH, Kupcinskas L, Kugathasan S, Latiano A, Laukens D, Lawrance IC, Lees CW, Louis E, Mahy G, Mansfield J, Morgan AR, Mowat C, Newman W, Palmieri O, Ponsioen CY, Potocnik U, Prescott NJ, Regueiro M, Rotter JI, Russell RK, Sanderson JD, Sans M, Satsangi J, Schreiber S, Simms LA, Sventoraityte J, Targan SR, Taylor KD, Tremelling M, Verspaget HW, De Vos M, Wijmenga C, Wilson DC, Winkelmann J, Xavier RJ, Zeissig S, Zhang B, Zhang CK, Zhao H; International IBD Genetics Consortium (IIBDGC); Silverberg MS, Annese V, Hakonarson H, Brant SR, Radford-Smith G, Mathew CG, Rioux JD, Schadt EE, Daly MJ, Franke A, Parkes M, Vermeire S, Barrett JC, Cho JH. Host-microbe interactions have shaped the genetic architecture of inflammatory bowel disease. Nature. 2012 Nov 1;491(7422):119-24. doi: 10.1038/nature11582. PMID 23128233